CLINICAL TRIAL: NCT05186506
Title: A Phase II, Open-Label, Randomized Study to Evaluate the Efficacy and Safety of Ensatinib Versus Platinum-Based Chemotherapy as Adjuvant Treatment for Stage II-IIIA ALK -Positive Non-Small Cell Lung Cancer
Brief Title: A Study Comparing Ensatinib Versus Platinum-Based Chemotherapy as Adjuvant Treatment for Stage II-IIIA ALK -Positive Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Collaborators: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Principal Investigator, You Lu, Chair of Department of Thoracic Oncology, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD-EN-IV005
Record Dates: First submitted 2021-12-29; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: ALK Fusion Protein Expression; Adjuvant Therapy; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ensartinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ensatinib (Experimental): 225 mg administered once daily orally for two years.
  Interventions: Drug: Ensatinib
- Platinum-Based Chemotherapy (Active Comparator): Patients in the chemotherapy group were allowed to cross into the Ensatinib treatment group after the disease progressed.
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Drug: Ensatinib — 225 mg administered once daily orally for two years.
  Other Names: X-396
  Arms: Ensatinib
Drug: chemotherapy — Pemetrexed : Participants will receive 500 mg/m^2, day 1 , Q21D , until completion of treatment period (4 cycles), recurrence of disease, unacceptable toxicity, withdrawal of consent, or death, whichever occurs first.
  Cisplatin :Participants will receive 75 mg/m^2, day 1 , 21 days/cycle, Q21D , until completion of treatment period (4 cycles), recurrence of disease, unacceptable toxicity, withdrawal of consent, or death, whichever occurs first.
  Paclitaxel: Participants will receive 175 mg/ m^2, day 1 , 21 days/cycle, Q21D , until completion of treatment period (4 cycles), recurrence of disease, unacceptable toxicity, withdrawal of consent, or death, whichever occurs first.
  carboplatin AUC= 5 mg/ mL/min, intravenously guttae, day 1 ,Q21D ，until completion of treatment period (4 cycles), recurrence of disease, unacceptable toxicity, withdrawal of consent, or death, whichever occurs first.
  Arms: Platinum-Based Chemotherapy

SUMMARY:
This randomized, active-controlled, multicenter, open-label, Phase II study is designed to evaluate the efficacy and safety of ensatinib compared with Platinum-Based Chemotherapy as adjuvant treatment in ALK fusion positive II-IIIA stage non-small cell lung cancer after surgical resection

DETAILED DESCRIPTION:
Participants in the experimental arm will receive Ensatinib at 225 mg orally once a day (QD) taken with food for 2 years. Participants in the control arm will receive one of the protocol specified platinum based chemotherapy regimens for 4 cycles. Treatments will continue until disease recurrence, meeting one of treatment discontinuation criteria (eg, patient decision, adverse event, pregnancy), or achieving a maximum treatment duration of 2 years. At the time of disease recurrence, participants will enter a survival follow-up until death, withdrawal of consent or study closure, whichever occurs earlier.

ELIGIBILITY:
Inclusion Criteria:

* Surgical resection of histologically confirmed Stage IIA to IIIA NSCLC with negative margins, ,within 10 weeks after the operation
* Documented ALK-positive disease according to FISH , Ventana IHC ,RT-PCR or NGS
* Eastern Cooperative Group (ECOG) Performance Status score of 0 or 1
* At least 3-months life expectancy
* Adequate organ function
* Any major surgery should be completed at least 4 weeks before the first study drug treatment. Minor surgery/procedures must be completed at least 2 weeks before taking medication.
* Willingness and ability to comply with the trial and follow-up procedures
* Written informed consents are required to indicate that the patients are aware of the investigational nature of the study

Exclusion Criteria:

* More than 10 weeks before surgery Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Use of other investigational drug within 4 weeks prior to the first dose of Ensartinib
* Prior stem cell or organ transplant
* severe cardiovascular disease
* Presence of active gastrointestinal (GI) disease or other conditions that will interfere significantly with the absorption, distribution, metabolism, or excretion of Ensartinib
* Active hepatitis B, hepatitis C virus antibody positive, HIV virus antibody, Treponema pallidum antibody positive
* History of interstitial lung disease, drug-induced interstitial lung disease, history of radiation pneumonitis requiring steroid therapy, or any clinical signs of active interstitial lung disease
* Reproductive or pregnant or breastfeeding female with a positive serum pregnancy test 7 days before starting treatment , Male or female patients failure to take effective contraceptive measures or plan to give birth during the entire treatment period and 3 months after treatment ends
* Patients with a known allergy or delayed hypersensitivity reaction to drugs chemically related to ensartinib or to the active ingredient of ensartinib
* History of drug allergy, such as a history of allergies to pemetrexed, carboplatin or other platinum compounds, or their preventive medications; History of allergies to paclitaxel components; or uncontrolled asthma
* Patients who have used the following drugs within 14 days before the first dose or who need to use the following drugs during treatment: drugs that cause QTc prolongation and/or torsade de pointes-type ventricular tachycardia; strong inhibitors or strong inducers of CYP3A
* Patients being treated with warfarin or any other coumarin derivative anticoagulant
* According to the judgment of the investigator, other severe, acute or chronic medical conditions that may increase the risk associated with participating in the study, or may interfere with the interpretation of the study results
* Concurrent condition evaluated by investigator that would make it inappropriate for the patient to be enrolled

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | From date of randomization until date of the first observation of tumor recurrence, metastasis (based on imaging ) or death, up to approximately 5 years.

SECONDARY OUTCOMES:
DFS at 2 years | Assessed at 2 years
DFS at 3 years | Assessed at 3 years
Overall survival (OS) | The time from the date of randomization to death from any cause, up to approximately 7 years
OS rate at 5 years | Assessed at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Study Chair — Sichuan University; Meijuan Huang, MD, Study Chair — Sichuan University

IPD SHARING:
Plan to Share IPD: No